CLINICAL TRIAL: NCT03661359
Title: Patient Perceptions of Care: The Effects of Social Determinants of Health
Brief Title: Social Determinants of Health Screening and Interventions
Acronym: SDOH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Sponsor
Organization: University of Toledo (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SDOH Study
Record Dates: First submitted 2018-06-20; First posted 2018-09-07 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Social Determinants of Health; Patient Satisfaction; Quality of Life
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Each patient who consents will be given the community resource interventions which apply to them based on the results of the Social Determinants of Health Screening Tool.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Social Determinants of Health (Experimental): Intervention will be the Social Determinants of Health Referrals.
  Interventions: Other: Social Determinants of Health Referrals

INTERVENTIONS:
Other: Social Determinants of Health Referrals — Patients who screen positive for any of the Social Determinants of Health will be given information for referral to any of the community resources that apply to their situation.

SUMMARY:
The primary objective of this study is to connect patients with community resources to improve social determinants of health. Secondary objectives are improving patient satisfaction within the trauma and general surgery service, enhancement of physician-patient communication, betterment of surgery department Hospital Consumer Assessment of Healthcare Providers and Systems scores, and increased understanding of correlations between patient satisfaction and social determinants of health.

The investigators hypothesize that (1) directed screening and intervention can have a positive effect for patients and hospitals, (2) directed patient advocacy will have an effect on patients' perception of care, (2) social determinants of health will have an effect on patients' perception of care, and (4) traumatic injury and acute surgery will have an effect on patients' perception of care.

DETAILED DESCRIPTION:
The investigators will be conducting this study as a prospective, non-randomized quality improvement study that will look at patients 18 years of age and older who are admitted under the trauma and general surgery specialties. Patients will be identified through admission to the trauma or general surgery service or referred to surgery services.

Eligible patients will be identified and approached by the study team. Once the informed consent is completed, patients will be given a Social Determinants of Health Screening Tool, an Hospital Consumer Assessment of Healthcare Providers and Systems Feedback Tool, and an short form health survey (SF-12) Quality of Life Questionnaire. Feedback from the Hospital Consumer Assessment of Healthcare Providers and Systems results will be given immediately to the relevant teams (nurses, doctors, etc.) to address the patient's concerns. Prior to discharge, the patients will also be given referrals to designated community resources. On day 15 (+/- 7 days) after discharge, the patients will receive a follow up phone call where they will be asked if they have utilized the Social Determinants of Health Referrals. Participants will also be given a second Hospital Consumer Assessment of Healthcare Providers and Systems Feedback Survey at this time. On day 30 (+/- 7 days) after discharge, the patients will receive a follow up phone call where the participants will be asked if they utilized the Social Determinants of Health Referrals. Participants will also be given a second short form health survey (SF-12) Quality of Life Survey at this time.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Admitted to the trauma or general surgery services
* Live within Lucas County (for county referrals)
* Patient or legally authorized representative agrees to participate and is willing to sign informed consent

Exclusion Criteria:

* Anyone less than 18 years old
* Any patient or legally authorized representative unwilling to sign informed consent
* Anyone who lives outside of Lucas County or expresses unwillingness to use referral services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Klepacz, MD, Principal Investigator — University of Toledo
Locations (1):
- University of Toledo Medical Center, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Data collection is still in early stages. Further discussion will be needed before a decision is finalized.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Social Determinants of Health
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Social Determinants of Health
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 8
Age, Continuous [Mean (Full Range); unit: years] | 44.97 [18 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Correlation Co-efficient Between Patient Satisfaction Assessed Using HCAHPS and the Domains at Risk
Description: evaluation of patient satisfaction of hospital and staff by patient questionnaire, abbreviated hospital consumer assessment of healthcare providers and system HCAHPS, 9 questions based on positive or negative patient response to hospital care. positive (yes) responses correlate to a 1, negative (no ) responses correlate to a 2. the lower the number correlates to higher hospital satisfaction score. also included a hospital rating of 1-10 with 1 being lowest score and 10 being the highest rating. A higher score correlates to a higher patient satisfaction level. Domains at risk related to social determinants of health
Time Frame: Within 15 days of discharge
Measure: Number; unit: correlation coefficient
Arm/Group | Social Determinants of Health
Number analyzed (Participants) | 35
correlation coefficient | -0.061
Statistical Analysis 1: Comparison: Social Determinants of Health; Correlation between patient satisfaction and domains at risk; Test type: Other; p = .727, pearson correlation — correlation is significant at the 0.05 level (2 tailed)

2. Primary Outcome: Patients Who Filled Out Community Service Questionnaires
Description: During hospital admission each consented patient was assessed for the 5 domains of social determinants of health. Domains are education, economic stability, environment, health/healthcare, and social/community with 11 questions including financial strain, food insecurity, training/employment, housing instability education, utility needs, transportation, childcare, exposure to violence, social connection, behavioral health/substance abuse. A positive (yes) response flagged the patient for a referral to a community service including community financial resources, food banks and kitchens, community employment and training programs, local shelters. adult education programs, utility assistance programs, community transportation programs, community day resources, domestic violence programs, community centers including senior and religious, mental health and substance abuse resources.
Time Frame: Within 30 days of discharge
Population: only 1 patient utilized the community resources available after discharge
Measure: Number; unit: participants
Arm/Group | Social Determinants of Health
Number analyzed (Participants) | 35
participants | 1

3. Primary Outcome: Correlation Co-efficient Between Physical Quality of Life and Mental Quality of Life
Description: evaluate the patients perception of their own health with a short form health questionnaire (SF-12).
  Physical component score (PCS-12): A score of 50 or less may indicate a physical condition.
  Mental component score (MCS-12): A score of 42 or less may indicate clinical depression.
  General health: Scores above 50 indicate better-than-average health, while scores below 50 indicate below-average health.
  This compares the physical and mental scores. A correlation coefficient is a statistical measure that indicates the strength and direction of a linear relationship between two variables, expressed as a number between -1 and 1, where -1 signifies a perfect negative correlation, 0 indicates no correlation, and +1 represents a perfect positive correlation; essentially, it tells you how closely two variables are related to each other in a linear fashion.
Time Frame: within 30 days of discharge
Measure: Number; unit: correlation coefficient
Arm/Group | Social Determinants of Health
Number analyzed (Participants) | 35
correlation coefficient | 0.5
Statistical Analysis 1: Comparison: Social Determinants of Health; correlation between physical quality of life and mental of life; Test type: Other; p = 0.002, pearson correlation — correlation is significant at the 0.01 level 2 tailed

4. Secondary Outcome: Communication Between Patient and Health Care Givers Questionnaire
Description: patients will evaluate the communication of the hospital staff with an abbreviated hospital consumer assessment of healthcare providers and system (HCAHPS) and rate the communication. the scale is based on positive (yes) or negative (no) responses. positive (yes) correlates to 1, negative (no) correlates to a 2. This scale of total answers can range from 1 to 10. One being the worst score and 10 being the best score. Once the questionnaire was completed. The negative (no) responses are shared with hospital leadership and unit directors to improve patient/staff communication.
Time Frame: Within 15 days of discharge
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | Social Determinants of Health
Number analyzed (Participants) | 35
Scores on a scale | 8 [1 to 10]

5. Secondary Outcome: Baseline HCAHPS Data
Description: Baseline data obtained for evaluation of patient satisfaction of hospital and staff by patient questionnaire, abbreviated hospital consumer assessment of healthcare providers and systems, HCAHPS. 10 questions total. 9 based on positive (yes) and negative (no) answers. Positive response (yes) correlates to number 1. negative response (no) correlates to a number 2. The lower the score the greater the patient satisfaction with the hospital. 1 question was a hospital rating scale of 1-10 with 1 being the lowest score and 10 being the highest score. A higher score correlates to a higher patient satisfaction level. A correlation coefficient is a statistical measure that indicates the strength and direction of a linear relationship between two variables, expressed as a number between -1 and 1, where -1 signifies a perfect negative correlation, 0 indicates no correlation, and +1 represents a perfect positive correlation; essentially, it tells you how closely two variables are related to ea
Time Frame: Within 15 days of discharge
Measure: Number; unit: correlation coefficient
Arm/Group | Social Determinants of Health
Number analyzed (Participants) | 35
correlation coefficient | -0.061
Statistical Analysis 1: Comparison: Social Determinants of Health; Test type: Other; p = 0.727, pearson correlation

ADVERSE EVENTS:
Time Frame: 37days
Arm/Group | Social Determinants of Health
All-Cause Mortality (participants affected / at risk) | 2/35
Serious Adverse Events (participants affected / at risk) | 2/35
Other Adverse Events (participants affected / at risk) | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Social Determinants of Health (N=35)
death (Injury, poisoning and procedural complications) | 1 (1) — patient was a victim of a violent crime
death (Social circumstances) | 1 (1) — patient died at home

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/59/NCT03661359/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/59/NCT03661359/ICF_001.pdf